CLINICAL TRIAL: NCT06896812
Title: A Pilot Study on App-based Treatment Combining Physical Exercise, Graded Activity, and Pain Journaling for Patients with Spinal Complaints
Acronym: SPINAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: The eHealth Project B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z2024093
Record Dates: First submitted 2025-03-06; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Back Pain; Spinal Disease; Spinal Condition
Keywords: conservative; app; spine; ehealth; e-health; back pain; graded activity
MeSH Terms: conditions — Back Pain; Spinal Diseases; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Study design: Single center prospective study.
  Study population: A total of 30 patients over 18 years old suffering from spinal complaints for which in current practice physical therapy, general lifestyle advice, or an expectant treatment will be advised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- App-based treatment consisting of physical exercise, graded activity, and pain journaling (Experimental): An app-based treatment consisting of a combination of physical exercise, graded activity, and pain journaling.
  Interventions: Device: The app-based treatment consists of a combination of physical exercise, graded activity, and pain journaling.

INTERVENTIONS:
Device: The app-based treatment consists of a combination of physical exercise, graded activity, and pain journaling. — The app-based treatment consists of a combination of physical exercise, graded activity, and pain journaling. The app will be installed on the participant's mobile device. The app will be used anonymously, and patients use their unique study code to activate the app.
  The content and user-interface of the app-based treatment were developed in collaboration with healthcare professionals for relevant medical specialties, including orthopedic surgery, neurosurgery, neurology, physiotherapy, and rehabilitation. The content is based on expert opinion from these fields. Additionally, there is scientific evidence indicating that the treatments used within the app are safe and effective. The app has been tested for usability and functionality by both professionals and laypersons, including individuals with back pain.

SUMMARY:
Background: The prevalence of spinal complaints such as low back pain is rising due to factors like aging, sedentary lifestyle, and obesity. Traditional conservative treatments include physical therapy and lifestyle modifications. The digital revolution in healthcare has introduced app-based interventions as a promising alternative.

Rationale: Given the high burden of spinal complaints and the associated economic impact, there is need for effective and efficient treatment modalities. This is especially evident in Western healthcare systems with growing demands and limited resources due to the changing demographic of the population. An app-based approach offers a viable solution by combining evidence-based conservative treatments. Moreover, an app-based treatment could offer personalized treatment, real-time feedback, and enhanced patient engagement at lower costs, presents as a viable solution.

Objective: This pilot study aims to evaluate the efficacy of an app-based treatment method combining physical exercise, graded activity, and pain journaling for patients with spinal complaints who will otherwise receive physical therapy, general lifestyle advice, or an expectant treatment in current practice.

Study design: Single center prospective study.

Study population: A total of 30 patients over 18 years old suffering from spinal complaints for which in current practice physical therapy, general lifestyle advice, or an expectant treatment will be advised.

Intervention: An app-based treatment consisting of a combination of physical exercise, graded activity, and pain journaling.

Main study parameters/endpoints: Primary endpoint: Patients' experience and satisfaction qualitatively, measured using semi-structured face-to-face interviews after three months of treatment.

Secondary endpoints: Quality of Life (Qol) measured with the EuroQol 5 dimensions (EQ-5D-5L) at baseline, one, two and three months after starting the intervention. Change in back- and leg-pain, measured with the Visual Analogue Scale (VAS). Change in disability, measured with the Oswestry Disability Index (ODI). Change in catastrophizing of pain, measured with the Pain Catastrophizing Scale (PCS). Change in lost productivity, measured with patient reported missed working days. Healthcare consumption, measured with number of visits to doctor or paramedic. Change in Body Mass Index, measured using patients' input on length and weight. Adherence of participants measured using frequency of patients' input in the mobile application. Safety measured using the (serious) adverse events ((S)AE).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The nature and extent of the burden associated with participation in the app-based treatment program primarily involve adherence to recommended activities and inputting relevant health data. Given that the investigators are integrating existing treatment modalities, such as physical exercise, graded activity, and pain journaling, the risks associated with participation are minimal, as these interventions are already deemed safe and widely practiced. The responsibility for determining each patient's suitability for participation in this study lies with the referring physician. Participants can expect benefits such as improved pain management, enhanced physical function, and better overall well-being.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   The incidence of spinal complaints is increasing in the ageing population. Back pain is amongst the conditions with the highest burden of disease in terms of years lived with disability (YLD), with a global lifetime prevalence of about 80%. The global prevalence of spine-related complaints is 9.4%, and this increases with age, reaching 19-23% by the age of 80. Besides age, spine-related disorders are also associated with a sedentary lifestyle and obesity. Consequently, as the population ages and rates of obesity and physical inactivity increase, the number of patients with spine-related disorders is rising exponentially. Besides causing significant pain and impairment, spinal complaints also impose an economic burden on healthcare systems worldwide. This economic burden is reflected by considerable healthcare-related costs and indirect costs such as loss of productivity.

   Traditional conservative interventions, such as physical therapy, pharmacological management, and lifestyle modifications are the most widely used modes of treatment for most spinal complaints, mainly back pain. It should be noted that there is conflicting evidence on the effect of most of these treatments, although there might be evidence for their effectiveness in the short term. It is apparent that physical therapy and lifestyle modifications focused on physical activity are the most successful options to achieve long term results.

   The digital revolution in the healthcare sector, characterized by rapid proliferation of health apps, offers promising avenues for innovative treatment modalities. These app-based interventions have potential to deliver personalized treatment regimens, provide real-time feedback, and enhance patient engagement, from the convenience of a patient's mobile device. Another possible benefit of app-based treatments is the wide availability and scalability at relatively low costs, especially when compared to traditional treatments.

   While these digital tools hold promise, there remains a critical need to assess their efficacy. Studies of healthcare apps in other fields have shown mixed results, with most indicating promising outcomes from app-based interventions, while some suggest only small benefits, like traditional treatment modalities.

   The challenges highlighted above are also evident in daily clinical practice. Clinicians frequently encounter patients with spine-related complaints that do not require a specific treatment. In current practice, these patients are referred to the general practitioner with general lifestyle advice, advise on physical activity management, and sometimes physical therapy. The exact advice is often based on the physicians' preferences. The vast majority of these patients is not followed up by the physician, and data on the effectiveness of the general advise is thus lacking.

   The investigators believe that an app-based treatment could address some of these barriers and provide meaningful support for a portion of the patient population. By offering standardized advice and guidance and fostering engagement through a convenient digital tool, an app-based interventions may empower patients to actively participate in their care. Moreover, a more standardized advice enables evaluation of the intervention. This study thus seeks to provide a comprehensive evaluation of the feasibility and efficacy of an app-based treatment for spinal complaints that do not require a specific intervention.
2. OBJECTIVES

Primary Objective:

To investigate the viability, feasibility, effectiveness, and safety of an app-based treatment combining physical exercise, graded activity, and pain journaling, by evaluating the patients' experience and satisfaction qualitatively, using semi-structured face-to-face interviews at three months follow-up in patients with spinal complaints who would receive physical therapy, general lifestyle advice, or an expectant treatment in current practice.

Secondary Objectives:

1. To assess change in quality of life, measured with the EuroQol 5 dimensions (EQ-5D-5L).
2. To assess the change in pain, measured with the Visual Analogue Scale (VAS).
3. To assess the change in disability, measured with the Oswestry Disability Index (ODI).
4. To assess the change in catastrophizing of pain, measured with the Pain Catastrophizing Scale (PCS).
5. To assess the change in lost productivity, measured with missed working days.
6. To assess healthcare consumption, measured in number of visits to doctor or paramedic.
7. To assess change in Body Mass Index, measured using patients' input on length and weight.
8. To evaluate the adherence of participants, measured using frequency of patients' input in the mobile application.
9. To evaluate the safety of the intervention, measured based on the occurrence of (serious) adverse events. Adverse events reported spontaneously by the subject or observed by the investigator or medical staff will be recorded.

Hypothesis:

An app-based treatment combining physical exercise, graded activity, and pain journaling is an effective, safe and feasible treatment option for the studied population.

3. STUDY DESIGN

A prospective pilot study with a treatment and follow-up duration of three months will be conducted in Zuyderland Medical Centre Heerlen, the Netherlands. The follow-up period of three months is chosen, as it is deemed appropriate to allow for a comprehensive evaluation of the app's usability, acceptance, and initial efficacy in managing spinal complaints. Moreover, a short study period reduces recall bias in qualitative data. A longer follow-up period, e.g. one year, would provide more data on long-term effects, but is beyond the scope of this pilot study.

This study includes patients with spinal complaints who would receive physical exercise, general lifestyle advice, or an expectant treatment, in current practice and do not require another specific treatment or surgical intervention. Patients eligible for inclusion will be referred to the researchers. The researchers will inform the patient, and when they are willing to participate and meet the inclusion criteria, include them. Patients will provide informed consent when first logging into the treatment app.

4. STUDY POPULATION 4.1 Population (base) Adult patients referred to the secondary spine-centre outpatient clinic suffering from spinal complaints are eligible to participate in the study. The treating clinicians will inform patients about the study. If patients are interested in participating, the patient will be referred to the researchers and receive the study information in writing. The researcher will then further inform the patient about the study verbally, and answer any remaining questions. The responsibility for determining each patient's suitability for participation in this study lies with the referring physician. The physician will evaluate whether the patient can safely engage with the app-based interventions, taking into account individual medical history, physical health, and any contraindications to physical activity. This evaluation ensures that each participant's medical needs and limitations are considered prior to inclusion, thereby supporting safe and effective use of the app's exercise recommendations.

4.2 Inclusion criteria

* Patients visiting the spine-centre at Zuyderland Medical Centre.
* Suffering from spinal complaints for which in current practice physical therapy, general lifestyle advice, or an expectant treatment would be advised.
* Minimum age of 18 years.
* Psychosocially, mentally, and physically able to fully comply with this study protocol.
* Informed consent prior to this study.

4.3 Exclusion criteria

* Requiring a specific intervention (e.g., surgery, pain treatment, rehabilitation, bracing)
* Inadequate command of the Dutch language.
* Digitally illiterate or otherwise unable to use an application on a mobile phone.
* Active spinal infection.
* Immature bone (ongoing growth).
* Active malignancy.
* Pregnancy.

4.4 Sample size calculation This study seeks to include 30 patients. This sample size has been chosen to allow for a comprehensive evaluation of the app's usability, acceptance, and initial efficacy in managing spinal complaints. By engaging this cohort, the investigators aim to gather valuable insights to determining the feasibility of proceeding with a larger-scale clinical trial. Additionally, findings derived from this group will allow adjustments and refinements to the app's functionalities.

5. TREATMENT OF SUBJECTS 5.1 Investigational product/treatment The app-based treatment consists of a combination of physical exercise, graded activity, and pain journaling. The app will be installed on the participant's mobile device. The app will be used anonymously, and patients use their unique study code to activate the app.

The content and user-interface of the app-based treatment were developed in collaboration with healthcare professionals for relevant medical specialties, including orthopedic surgery, neurosurgery, neurology, physiotherapy, and rehabilitation. The content is based on expert opinion from these fields. Additionally, there is scientific evidence indicating that the treatments used within the app are safe and effective. The app has been tested for usability and functionality by both professionals and laypersons, including individuals with back pain. Based on the experience of the involved professionals, it was decided not to include muscle-strengthening exercises in the app. This decision was made because, for some patients, muscle-strengthening exercises may be overly strenuous without contributing to recovery, and they may even have counterproductive effects. Furthermore, as these exercises are performed without the direct supervision or control of a physical therapist, including muscle-strengthening exercises would have too great an impact on the "one-size-fits-most" design of the study.

Physical exercise

Patients are instructed to perform several stretches daily. It is advised to perform each stretch for 20-30 seconds. Patients will receive information on how to properly perform these stretches through text, images, and optional videos. The included stretches are:

1. Cat-cow stretch or a combination of pelvic tilts and knees to chest stretch.
2. Seated or standing hamstring stretch.
3. Kneeling or standing hip flexor stretch.
4. Seated or lying thoracic rotations.

Graded activity In the graded activity section of the app, patients chose either walking or bicycling, based on their own preferences. Both graded activity programs have the same structure. The program starts with a baseline self-assessment. Patients determine how many minutes they can perform the activity before the pain reaches VAS 7 (significant pain). This number of minutes is then applied in the graded activity program. Pain scores are monitored during and after activity.

Frequency: Once every day. If the duration of the activity exceeds 10 minutes, the frequency is adjusted to once every two days.

Duration: Start with a duration that 70% of the baseline assessment. For instance, if the patient can walk for 10 minutes before pain intensifies to a level at which the patient has to stop, start with 7 minutes.

Pain Score Monitoring: If the planned activity is not reached due to pain, the duration of activity is not adjusted.

Incremental Increase: Increase the duration by 10% after each activity without significant pain, with a minimal increase of one minute.

Steady State: If the patient is able to walk for longer than half an hour without significant pain, no adjustments are made.

Pain Journaling

The app incorporates pain and symptom journaling. The app uses graphics to provide patients with insight on the symptoms, exercise frequency and activity. The following components are included:

1. Daily: Exercises logging, VAS back pain score & analgesics used (paracetamol, NSAIDs, opioids, neuropathic analgesics, other).
2. Seven - three times a week, depending on level of activity: activity (minutes) and VAS back pain during and after activity.
3. Monthly: Health-related quality of life (EQ-5D-5L), disability (Oswestry Disability Index), pain catastrophizing (PCS), weight (kilograms), work absenteeism (days, including unpaid work), healthcare consumption (number of visits to doctor or paramedic).

5.2 Use of co-intervention There will be no specific co-interventions. Use of analgesia is continued or adjusted based on the advice of the general practitioner or treating medical doctor, no adjustment will be suggested by the app. Although patients are not actively advised to seek additional treatment, patients are allowed to seek additional treatment or support from paramedical professionals on their own initiative if desired. This may include visits to physical therapists, chiropractors, acupuncturists, or other healthcare providers for supplementary treatment or guidance. These options allow participants to pursue complementary therapies alongside the app-based program, should they feel that additional support aligns with their personal recovery goals and preferences. Patient reported healthcare consumption will be assessed as part of this study. Moreover, co-interventions will be evaluated qualitatively during the interviews.

6. INVESTIGATIONAL PRODUCT

6.1 Name and description of investigational product(s) Rug App (as developed by The eHealth Project B.V.) 6.2 Summary of findings from non-clinical studies None. 6.3 Summary of findings from clinical studies None. 6.4 Summary of known and potential risks and benefits None. 6.5 Description and justification of route of administration and dosage Not applicable. 6.6 Dosages, dosage modifications and method of administration Not applicable. 6.7 Preparation and labelling of Investigational Medicinal Product Not applicable. 6.8 Drug accountability Not applicable.

8. METHODS 8.1 Study parameters/endpoints 8.1.1 Main study parameter/endpoint The primary outcome is qualitative information on the viability, feasibility, effectiveness, and safety. The data used is gathered by evaluating the patients' experience and satisfaction qualitatively, using semi-structured face-to-face interviews at three months follow-up.

8.1.2 Secondary study parameters/endpoints

* Demographics
* Cange in QoL, measured with the ED-5D-5L.
* Change in pain, measured with the Visual Analogue Scale (VAS).
* Change in disability, measured with the Oswestry Disability Index (ODI).
* Change in lost productivity, measured with missed working days.
* Change in Body Mass Index, measured using patients' input on length and weight.
* Healthcare consumption, measured in number of visits to doctor or paramedic.
* Adherence of participants measured using frequency of patients' input in the mobile application.
* Safety measured using the (serious) adverse events ((S)AE).

Adverse events: increased pain or discomfort for which the patient visits the hospital, neurological deficits, technology-related issues. Adverse events will be followed up to 30 days after completion of the treatment period.

8.2 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

9. SAFETY REPORTING 9.1 Temporary halt for reasons of subject safety In accordance with section 10, subsection 4, of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardize subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

9.2 AEs, SAEs and SUSARs 9.2.1 Adverse events (AEs) Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the experimental intervention. All adverse events reported spontaneously by the subject or observed by the investigator, or his staff will be recorded. This also includes the described complications such increased pain or discomfort for which the patient visits the hospital, neurological deficits, technology-related issues.

9.2.2 Serious adverse events (SAEs) A serious adverse event is any untoward medical occurrence or effect that

* results in death.
* is life threatening (at the time of the event).
* requires hospitalization or prolongation of existing inpatients' hospitalization.
* results in persistent or significant disability or incapacity.
* is a congenital anomaly or birth defect; or
* any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator. This also includes the described complications such as postoperative infection, deep venous thrombosis, hematoma, neurological deficits and other complications as pneumonia, urine retention or urinary tract infection.

An elective hospital admission will not be considered as a serious adverse event.

The investigator will report all SAEs to the sponsor without undue delay after obtaining knowledge of the events.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

9.2.3 Suspected unexpected serious adverse reactions (SUSARs) The investigator will report all SUSARs to the sponsor within 15 days of obtaining knowledge of the events. The sponsor will report these SUSARs to the accredited METC every six months.

10. ETHICAL CONSIDERATIONS 10.1 Regulation statement This research will be conducted according to the principles enshrined in the Declaration of Helsinki (7th edition 2013) and in accordance with the Medical Research Involving Human Subjects Act (WMO, version 1 July 2012).

10.2 Recruitment and consent Adult patients referred to the secondary spine-center outpatient clinic suffering from spinal complaints for which in current practice physical therapy, general lifestyle advice, or an expectant treatment would be advised are eligible to participate in the study and will be referred by colleagues to the researchers. Patients who are interested in participating in this study will receive the study information orally by their physician and in writing, along with the patient information. When a patient is informed about the study and considers participating in the study, the patient receives a unique study code (e.g., Z01, Z02, Z02, etc.), along with a code-specific password that is needed to access the content of the app. The informing doctor or researcher notifies the principal investigator which patient received which unique code. The app is not accessible until the patient digitally signs the informed consent.

After one week, researchers will call the patient to check if they have any more questions and want to participate. If patients want to be included in the study, they can sign the informed consent in the app using their unique, pseudonymized login credentials. On the informed consent page of the app, all study information is digitally available to the patients.

Identification, authentication, and authorization are warranted by means of these unique and patient-specific login credentials combined with telephone contact by the researcher prior to study participation. Patients will receive a signed and dated copy if the informed consent form by mail.

After inclusion of the participant, he/she has the right to always terminate his participation, without giving reasons. Participation can be terminated by the patients in the settings of the app. In this case standard treatment will be continued. For any questions regarding the study, an independent physician is available for the duration of the study. If the patient chooses not to participate in the study, standard treatment will be offered.

Additional information about handling and storage of data can be found in chapter 12 and the Funding Agreement.

11.3 Objection by minors or incapacitated subjects (if applicable) Not applicable.

10.4 Benefits and risks assessment, group relatedness The nature and extent of the burden associated with participation in the app-based treatment program primarily involve adherence to the recommended activities and inputting relevant health data. Adherence to the prescribed activity and inputting data will take several minutes per day. Based on tolerance to activity, this may amount to a maximum of three hours per week. Given that the investigators are integrating existing treatment modalities such as physical exercise, graded activity, and pain journaling, the risks associated with participation are minimal, as these interventions are already deemed safe and widely practiced.

The responsibility for determining each patient's suitability for participation in this study lies with the referring physician. The physician will evaluate whether the patient can safely engage with the app-based interventions, taking into account individual medical history, physical health, and any contraindications to physical activity. This evaluation ensures that each participant's medical needs and limitations are considered prior to inclusion, thereby supporting safe and effective use of the app's exercise recommendations.

Participants can expect benefits such as improved pain management, enhanced physical function, and better overall well-being. Additional educational information such as frequently asked question and red flags included in the app are based on professional guidelines. Moreover, the application refers to professional and reliable information, specifically developed for Dutch patients (thuisarts.nl).

10.5 Compensation for injury The sponsor/investigator has a liability insurance which is in accordance with article 7 of the WMO. The sponsor (also) has an insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO). This insurance provides cover for damage to research subjects through injury or death caused by the study.

The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

10.6 Incentives Not applicable.

11. STRUCTURED RISK ANALYSIS 11.1 Potential issues of concern

1. Level of knowledge about mechanism of action Not applicable.
2. Previous exposure of human beings with the test product(s) and/or products with a similar biological mechanism.

   The specific app has not been tested yet. However, given that the investigators are integrating a combination of existing treatment modalities such as physical exercise, graded activity, and pain journaling, the risks associated with participation are minimal, as these interventions are already deemed safe and widely practiced results. Moreover, similar types of digital interventions are being developed and tested for patients suffering from low back pain and show promising results.
3. Can the primary or secondary mechanism be induced in animals and/or in ex-vivo human cell material? Not applicable.
4. Selectivity of the mechanism to target tissue in animals and/or human beings Not applicable.
5. Analysis of potential effect See point b. Serious adverse events or complications are not te be expected based on the type of intervention.
6. Pharmacokinetic considerations Not applicable.
7. Study population This study will only include adult patients with spinal complaints that do not require a specific treatment, such as surgery, bracing, etc.. Nor will this study include patients with active spinal infection, malignancy, pregnancy.
8. Interaction with other products Not applicable.
9. Predictability of effect As mentioned in point b., the effect and safety of treatment modalities used in the application are thoroughly investigated and well-know. Similar digital treatments show promising results. This ensures high predictability of the effect of the intervention.
10. Can effects be managed? In case of (serious) adverse events, medical support, and additional treatment in the outpatient clinic of at the emergency department is warranted.

11.2 Synthesis The nature and extent of the burden associated with participation in the app-based treatment program primarily involve adherence to recommended activities and inputting relevant health data. Given that the investigators are integrating existing treatment modalities such as physical exercise, graded activity, and pain journaling, the risks associated with participation are minimal, as these interventions are already deemed safe and widely practiced. Participants can expect benefits such as improved pain management, enhanced physical function, and better overall well-being. The risk of (serious) adverse events is low.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting the spine-centre at Zuyderland Medical Centre.
* Suffering from spinal complaints for which in current practice physical therapy, general lifestyle advice, or an expectant treatment would be advised.
* Minimum age of 18 years.
* Psychosocially, mentally, and physically able to fully comply with this study protocol.
* Informed consent prior to this study.

Exclusion Criteria:

* Requiring a specific intervention (e.g., surgery, pain treatment, rehabilitation, bracing)
* Inadequate command of the Dutch language.
* Digitally illiterate or otherwise unable to use an application on a mobile phone.
* Active spinal infection.
* Immature bone (ongoing growth).
* Active malignancy.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is qualitative information on the viability, feasibility, effectiveness, and safety. | 3 months
  The data used is gathered by evaluating the patients' experience and satisfaction qualitatively, using semi-structured face-to-face interviews at three months follow-up.

SECONDARY OUTCOMES:
Secondary outcome, Quality of Life | 3 months
  Change in QoL, measured with the ED-5D-5L.
Secondary outcome, pain | 3 months
  Change in pain, measured with the Visual Analogue Scale (VAS).
Secondary outcome, disablity | 3 months
  Change in disability, measured with the Oswestry Disability Index (ODI). o
Secondary outcome, productivity | 3 months
  Change in lost productivity, measured with missed working days.
Secondary outcome, BMI | 3 months
  Change in Body Mass Index, measured using patients' input on length and weight.
Secondary outcome, healthcare consumption | 3 months
  Healthcare consumption, measured in number of visits to doctor or paramedic.
Secondary outcome, adherence | 3 months
  Adherence of participants measured using frequency of patients' input in the mobile application.
Secondary outcome, safety | 3 months
  Safety measured using the (serious) adverse events ((S)AE).
  Adverse events: increased pain or discomfort for which the patient visits the hospital, neurological deficits, technology-related issues. Adverse events will be followed up to 30 days after completion of the treatment period.

IPD SHARING:
Plan to Share IPD: Undecided
Information about the study and access to anonymized data will be available on reasonable request.

REFERENCES:
- [Background] Nordstoga AL, Aasdahl L, Sandal LF, Dalager T, Kongsvold A, Mork PJ, Nilsen TIL. The Role of Pain Duration and Pain Intensity on the Effectiveness of App-Delivered Self-Management for Low Back Pain (selfBACK): Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Aug 31;11:e40422. doi: 10.2196/40422. PMID 37656023
- [Background] Bardal EM, Sandal LF, Nilsen TIL, Nicholl BI, Mork PJ, Sogaard K. Do age, gender, and education modify the effectiveness of app-delivered and tailored self-management support among adults with low back pain?-Secondary analysis of the selfBACK randomised controlled trial. PLOS Digit Health. 2023 Sep 22;2(9):e0000302. doi: 10.1371/journal.pdig.0000302. eCollection 2023 Sep. PMID 37738237
- [Background] Friese, S., Qualitative data analysis with ATLAS. ti. 2019.
- [Background] Hasenohrl T, Windschnurer T, Dorotka R, Ambrozy C, Crevenna R. Prescription of individual therapeutic exercises via smartphone app for patients suffering from non-specific back pain : A qualitative feasibility and quantitative pilot study. Wien Klin Wochenschr. 2020 Mar;132(5-6):115-123. doi: 10.1007/s00508-020-01616-x. Epub 2020 Feb 14. PMID 32060724
- [Background] Lau AY, Piper K, Bokor D, Martin P, Lau VS, Coiera E. Challenges During Implementation of a Patient-Facing Mobile App for Surgical Rehabilitation: Feasibility Study. JMIR Hum Factors. 2017 Dec 7;4(4):e31. doi: 10.2196/humanfactors.8096. PMID 29217504
- [Background] Meinert E, Rahman E, Potter A, Lawrence W, Van Velthoven M. Acceptability and Usability of the Mobile Digital Health App NoObesity for Families and Health Care Professionals: Protocol for a Feasibility Study. JMIR Res Protoc. 2020 Jul 22;9(7):e18068. doi: 10.2196/18068. PMID 32706703
- [Background] Sandal LF, Bach K, Overas CK, Svendsen MJ, Dalager T, Stejnicher Drongstrup Jensen J, Kongsvold A, Nordstoga AL, Bardal EM, Ashikhmin I, Wood K, Rasmussen CDN, Stochkendahl MJ, Nicholl BI, Wiratunga N, Cooper K, Hartvigsen J, Kjaer P, Sjogaard G, Nilsen TIL, Mair FS, Sogaard K, Mork PJ. Effectiveness of App-Delivered, Tailored Self-management Support for Adults With Lower Back Pain-Related Disability: A selfBACK Randomized Clinical Trial. JAMA Intern Med. 2021 Oct 1;181(10):1288-1296. doi: 10.1001/jamainternmed.2021.4097. PMID 34338710
- [Background] Snoswell CL, Chelberg G, De Guzman KR, Haydon HH, Thomas EE, Caffery LJ, Smith AC. The clinical effectiveness of telehealth: A systematic review of meta-analyses from 2010 to 2019. J Telemed Telecare. 2023 Oct;29(9):669-684. doi: 10.1177/1357633X211022907. Epub 2021 Jun 29. PMID 34184580
- [Background] Loohuis AMM, Van Der Worp H, Wessels NJ, Dekker JH, Slieker-Ten Hove MCP, Berger MY, Vermeulen KM, Blanker MH. Cost-effectiveness of an app-based treatment for urinary incontinence in comparison with care-as-usual in Dutch general practice: a pragmatic randomised controlled trial over 12 months. BJOG. 2022 Aug;129(9):1538-1545. doi: 10.1111/1471-0528.17191. Epub 2022 May 31. PMID 35460163
- [Background] Mahtta D, Daher M, Lee MT, Sayani S, Shishehbor M, Virani SS. Promise and Perils of Telehealth in the Current Era. Curr Cardiol Rep. 2021 Jul 16;23(9):115. doi: 10.1007/s11886-021-01544-w. PMID 34269884
- [Background] Krebs P, Duncan DT. Health App Use Among US Mobile Phone Owners: A National Survey. JMIR Mhealth Uhealth. 2015 Nov 4;3(4):e101. doi: 10.2196/mhealth.4924. PMID 26537656
- [Background] van Tulder MW, Koes BW, Bouter LM. Conservative treatment of acute and chronic nonspecific low back pain. A systematic review of randomized controlled trials of the most common interventions. Spine (Phila Pa 1976). 1997 Sep 15;22(18):2128-56. doi: 10.1097/00007632-199709150-00012. PMID 9322325
- [Background] Bredow J, Bloess K, Oppermann J, Boese CK, Lohrer L, Eysel P. [Conservative treatment of nonspecific, chronic low back pain : Evidence of the efficacy - a systematic literature review]. Orthopade. 2016 Jul;45(7):573-8. doi: 10.1007/s00132-016-3248-7. German. PMID 27075679
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Background] Weiner DK, Kim YS, Bonino P, Wang T. Low back pain in older adults: are we utilizing healthcare resources wisely? Pain Med. 2006 Mar-Apr;7(2):143-50. doi: 10.1111/j.1526-4637.2006.00112.x. PMID 16634727
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] Smith E, Hoy DG, Cross M, Vos T, Naghavi M, Buchbinder R, Woolf AD, March L. The global burden of other musculoskeletal disorders: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Aug;73(8):1462-9. doi: 10.1136/annrheumdis-2013-204680. Epub 2014 Mar 3. PMID 24590181
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116